CLINICAL TRIAL: NCT03559140
Title: Reduction of Post-endodontic Pain After Single-visit RCT Using Three Irrigating Regimens.
Brief Title: Reduction of Post-endodontic Pain After 3 Irrigation Regime
Acronym: RPEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, Chairman of Post graduate Programs in Dentistry, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: post endodontic pain 2018
Record Dates: First submitted 2018-04-22; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Post-operative Pain
Keywords: post-endodontic pain; pain; root canal treatment; cryotherapy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Random Selection of instrumentation groups. Of the sample of 216 teeth, 72 were randomly assigned to the one of the 3 irrigating methods. Treatment was performed by 3 experienced endodontists; each prepared 72 teeth, 24 per technique.
Who Masked: Participant, Investigator
Masking Description: Certified endodontists trained in the procedures, devices, and systems investigated took part in the research. All experts tracked a pre-established procedure for Reciproc instrument systems and cryotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): The R25 (size 25/ .08) instrument was used in thin and curved root canals, and R40 files (40/ .06) were used in wide root canals. Three in-and-out pecking motions were used with an amplitude of not more than 3 mm until reaching the estimated working length.
  After the procedure cryotherapy will be applied as follows:
  Patients assigned to this group receive a final irrigation (application of cryotherapy) with 5 mL cold (2.5oC) 17% EDTA followed with 20 mL cold (2.5oC) sterile saline solution delivered to the WL using a cold (2.5oC) sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes
  Interventions: Procedure: Applied saline solution at 8oC (Cryotherapy )
- Group B (Experimental): Canals were prepared as in group A, Patients assigned to this group receive (application of criotherapy)
  A final irrigation will be applied with 5 mL cold (2.5oC) 17% EDTA followed with 20 mL cold (2.5oC) sterile saline solution delivered to the WL using a cold (2.5oC) sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes. was applied. as follows:
  Patients assigned to this group receive a final irrigation (application of cryotherapy) with 5 mL cold (2.5oC) 17% EDTA followed with 20 mL cold (2.5oC) sterile saline solution delivered to the WL using a cold (2.5oC) sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes
  Interventions: Procedure: Applied saline solution at 2.5 oC (Cryotherapy group)
- Control Group (CG) (Experimental): The R25 (size 25/ .08) instrument was used in thin and curved root canals, and R40 files (40/ .06) were used in wide root canals. Three in-and-out pecking motions were used with an amplitude of not more than 3 mm until reaching the estimated working length. Reciproc instruments were used in one tooth only (single use).
  The group will receive the irrigant solution at room temperature. as follows:
  they will receive a final irrigation ( application of irrigant at room temperature) with 5 mL (room temperature) 17% EDTA followed with 20 mL (room temperature) sterile saline solution delivered to the WL using a sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes.
  Interventions: Procedure: Applied saline solution at room temperature (No cryotherapy)

INTERVENTIONS:
Procedure: Applied saline solution at 2.5 oC (Cryotherapy group) — Patients assigned to this group will receive a final irrigation (application of cryotherapy) with 5 mL cold (8oC) 17% EDTA followed with 20 mL cold (8oC) sterile saline solution delivered to the WL using a cold (8oC) sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes.
  Arms: Group B
Procedure: Applied saline solution at 8oC (Cryotherapy ) — Patients assigned to this group receive a final irrigation (application of cryotherapy) with 5 mL cold (2.5oC) 17% EDTA followed with 20 mL cold (2.5oC) sterile saline solution delivered to the WL using a cold (2.5oC) sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes.
  Arms: Group A
Procedure: Applied saline solution at room temperature (No cryotherapy) — Patients assigned to this control group were treated identically to the experimental groups, except that they will receive a final irrigation ( application of irrigant at room temperature) with 5 mL (room temperature) 17% EDTA followed with 20 mL (room temperature) sterile saline solution delivered to the WL using a sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes.
  Arms: Control Group (CG)

SUMMARY:
The goal of this research was to relate the occurrence of post-endodontic pain after single-visit RCT using there irrigating regime. Methodology: All 216 patients had upper or lower molar, premolar or anterior teeth selected for conventional RCT for prosthetic reasons detected with only vital pulps. Of the sample of 216 teeth, were selected to just one method for instrumentation and different manner to irrigate. All instruments were used with a micro motor (VDW, Munich Germany). Reciproc instruments. Final irrigation with cold (8oC, 2.5 oC and room temperature 17% EDTA and saline solution served as a lubricants.

DETAILED DESCRIPTION:
Two hundred and sixteen of 245 patients (119 women and 97 men) aged 18-65 years were referred and incorporated in this research while 29 were excluded as not meeting the inclusion criteria. All patients presented with a vital upper or lower molar, premolar or anterior teeth selected for conventional root canal treatment for prosthetic reasons.

Patients rejecting to join the study or rejecting, single-visit root canal treatment, consuming analgesics or NSAIDs were excluded too. All participants were informed on the goals, risks and strategy of the study, and written informed consent permissions were gained previous their enrollment.

Random Selection of instrumentation groups. An investigator who had not contributed in the study made the randomization arrangement using a computer random table generator (www.random.org). Each patient receive a consecutive number. A total of 216 patients met the inclusion requirements and were incorporated in the study. Of the sample of 216 teeth, 72 were randomly assigned to the one of the 3 irrigating methods. Treatment was performed by 3 experienced endodontists; each prepared 72 teeth, 24 per method.

Treatment Protocol All patients were anesthetized with two carpules of articaine 2% with epinephrine 1:200,000 (Septodont, Saint-Maur des-Fosses, France). In cases in which supplemental anesthesia was needed, intraligamental anesthesia (2 mL articaine 2%) was administered. For the upper teeth, the 2 carpules were administered by gradual infiltration in the buccal vestibule. For the lower teeth, 1.5 of the carpules was used for an inferior alveolar nerve block and the other 1.5 for a gentle buccal infiltration around the tooth to be treated.

After absolute isolation using rubber dam, the tooth was disinfected with 5.25% NaOCl. Preparation of the access cavity was performed using # 331 bur (Dentsply International, York, PA), with high-speed and water cooling. 5.25% NaOCl was used to clean the coronal cavity. The root canals were carefully probed with #10 K-type hand files (Flex-R files, Moyco/Union Broach, York PA, USA).

REDTA (Roth International, Chicago, IL) lubricant was located at the entry of the canals. Working length was determined with a #15 k-file and the Root ZX electronic device (J Morita, Irvine CA, USA), followed by subtracting 0.5 mm from the measurement, which was confirmed radiographically (Schick Technologies, NY, USA). Cervical and middle thirds of the root canal was flared with a K3XF 25/10 rotary instrument (Kerr Endo, Orange County, CA) at 500 rpm. The root canal was irrigated with 3 mL 5.25% sodium hypochlorite (NaOCl). A glide path to the WL was the established.

For mechanical preparations, all instruments were used with a micro motor (VDW Silver Motor, VDW, Munich Germany). Torque and rotation were preset for each Reciproc instrument. Rotary Ni-Ti instruments were used in continuous reciprocating mode.

Dentinal debris was eliminated from the file with a gauze, instantaneously to the instrument change after 2-3 in-and-out (pecking) movements (Reciproc) following the manufacturers' recommendations. Each root canal was irrigated with 2.5mL 2.6% NaOCl. Irrigation was performed using a 24-gauge needle (Max-I-Probe; Tulsa Dental, York, PA) and a 31-G NaviTip needle (Ultradent Products Inc, South Jordan, UT) when reaching the WL after each instrument insertion. A size #10 K file was used to maintain WL after each Reciproc instrument.

Group A. The R25 (size 25/ .08) instrument was used in thin and curved root canals, and R40 files (40/ .06) were used in wide root canals. Three in-and-out pecking motions were used with an amplitude of not more than 3 mm until reaching the estimated working length. Patients assigned to this group receive a final irrigation with 5 mL cold (8oC) 17% EDTA followed with 20 mL cold (8oC) sterile saline solution delivered to the WL using a cold (8oC) sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes.

Group B. Canals were prepared as in group A, Patients assigned to this group receive a final irrigation with 5 mL cold (2.5oC) 17% EDTA followed with 20 mL cold (2.5oC) sterile saline solution delivered to the WL using a cold (2.5oC) sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes.

Control group (CG). The R25 (size 25/ .08) instrument was used in thin and curved root canals, and R40 files (40/ .06) were used in wide root canals. Three in-and-out pecking motions were used with an amplitude of not more than 3 mm until reaching the estimated working length. Reciproc instruments were used in one tooth only (single use). Patients assigned to this control group were treated identically to the experimental groups, except that receive a final irrigation with 5 mL (room temperature) 17% EDTA followed with 20 mL (room temperature) sterile saline solution delivered to the WL using a sterile microcannula attached to the Endo Vac System (Kerr Endo) for 5 minutes.

After instrumentation, the root canals were irrigated with 1 mL 2.6% NaOCl, agitated ultrasonically. Ultrasonic activation was performed using an Irrisafe ultrasonic 20.00 tip (Satelec, Merignac, France) at 50% power of the MiniEndo ultrasonic unit (Kerr Endo) with the tip placed 3 mm from the working length for 30 seconds per root canal.

Each experimental and control group received a final irrigation with the irrigant described above, to eliminate the smear layer and reduce post-endodontic pain. Caution was taken to ensure that the micro cannula would suction correctly by detecting the system's transparent evacuation tube. In case there was any obstruction, the micro cannula was instantly substituted.

Recapitulation of working length was performed again by using an apex locator as described before using #35 and #40 files.

The root canals were dried with disinfected paper points and obturated at the same visit. Gutta-percha cones (Dentsply Maillefer) were laterally compacted with #20 nickel-titanium spreaders (Dentsply Maillefer) and AH-plus as the sealer (Dentsply Maillefer). The access cavities of anterior and posterior teeth were etched and repaired with Fuji IX (GC Corp, Tokyo, Japan).

Assessment of Post-endodontic pain and Statistical Analysis After these irrigation regimens, the patients were informed of the probable incidence of pain for days following RCT and received a survey form (VAS questionnaire) to be finished and returned three days after. In it, they proof the presence/absence of post-endodontic pain. The pain level was measured using a validated pain scale known as the VAS. The pain VAS is a continuous scale comprised of a horizontal line, which is 10 cm in length. For pain intensity, the VAS is anchored by ''no pain'' (score of 0) and ''pain as bad as it could be'' (score of 10). The cut points on the pain VAS are no pain (0-0.5 cm), mild pain (0.6-4.0 cm), moderate pain (0.45-7.4 cm), and severe pain (7.5-10 cm). The pain VAS was completed by the patients. The patients were asked to put a mark perpendicular to the pain VAS line at the point that indicated their pain severity during the 3 days after the endodontic treatment.

Two hundred and ten of the 216 surveys were returned correctly returned. Of these, 69 belonged to the group A, 70 to group B and 71 to the Control group. The missing 6 questionnaires were returned one day later and were included in the data analysis.

The outcomes for the groups A, B and CG associated to occurrence (yes/no), level (mild, moderate, severe), and interval (days) of post-endodontic pain were evaluated, and related to the following diagnostic factors: condition of tooth (all vital), occurrence or nonappearance of pre-operative pain, group of teeth (molar/premolar or anterior), or location (Maxillary, Mandibular).

ELIGIBILITY:
Inclusion Criteria:

* absence of radiographic sign of apical periodontitis and a diagnosis of irreversible pulpitis (IP) established by affirmative response to hot and cold examinations.

  * Thermal pulp examination was achieved by the corresponding author, and radiographic analysis was established by 3 certified endodontists.
  * Clinical requirements were established on the next conditions: 1) The purposes and necessities of the research were spontaneously accepted. 2) Clinical Management was pointed to patients in physical and mental well- being. 3) All teeth had vital pulps and absence of apical periodontitis. 4) Positive thermal stimulation with EndoIce (Hygenic Corp, Akron, OH). 5) Teeth with enough coronal structure for rubber dam isolation. 6) No RCT done before the research. 7) No painkillers or antibiotics used 7 days' prior the clinical events started

Exclusion Criteria:

* Exclusion parameters were:

  * the necessity for retreatment
  * gravidity
  * impossibility to obtain patient's approval
  * patients who didn't complete inclusion necessities
  * a history of medication for chronic pain or those compromising the immune response
  * patients younger than 18 years and the existence of mishaps or difficulties during RCT (calcified canals, impracticality of achieving AP in any can

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the post-endodontic pain after 24 hrs,48 and 72 hrs. | 24 hours to 72 hours
  Post-endodontic pain was evaluated after root canal treatment in order to identify in 216 patients: none, mild or severe pain.

SECONDARY OUTCOMES:
Evaluate the effect of intracanal cryotherapy on post-endodontic pain after root canal treatment. | 24 hours to 72 hours
  Post endodontic pain was evaluated after a final irrigation with cold 5cc of (2.5-8oC) 17% EDTA gently delivered to the WL using a cold (2.5-8oC) sterile metallic micro cannula.

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Paredes Vieyra, Tijuana, Baja Califronia, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729